CLINICAL TRIAL: NCT02879474
Title: Study of Risk Factors and Clinical Characterization of Rapidly Growing Melanoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: AORC 2009; RC13_0082 (Other: AP-HM)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with melanoma
  Interventions: Behavioral: Melanoma scale questionnair

INTERVENTIONS:
Behavioral: Melanoma scale questionnair

SUMMARY:
State of the question Over the past decade, the incidence of melanoma (MM) has steadily increased in France and in most developed countries. This increased incidence was concerned mainly MM thin while the incidence of MM thick that represent the true "killers", and mortality from MM remained stable or increased slightly over the same period. These epidemiological data and observations from everyday medical practice dermatologists suggest the existence of different growth patterns within MM. Indeed, some MM progressing slowly sometimes for decades before diagnosis but are thin at the time of resection. Conversely, others MM grow very quickly, resulting in thick tumors despite a diagnosis and resection sometimes very early. These fast growing MM (FGMM) probably contribute significantly to the relative mortality in MM, as improved screening failed to influence to this day.

Our team has already demonstrated that the growth kinetics of the MM was a prognostic factor of tumor aggressiveness regardless of the thickness of the tumor. Using the same method to calculate the growth rate, an Australian team recently studied the growth rate in a population of patients suffering from MM. In this population 1/3 of MM had a growth of more than 0.5 mm per month. Clinical aspects and FGMM of these risk factors were individuals (injuries symmetrical achromic and regular occurrence among about older and low-nevi). The European and Australian people are very different in particular regarding the prevention policy, these results can not be extrapolated to the French population.The main objective is to identify risk factors for FGMM in French propulation

ELIGIBILITY:
Inclusion Criteria:

* Patient with Breslow primitive melanoma for over 1 mm skin affected

Exclusion Criteria:

* Patient unable to answer questionnair concerning its melanoma history desease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breslow primitive melanoma >1 mm patients
Sampling Method: Probability Sample
Enrollment: 472 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Speed growth of melanoma size | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; Caroline GAUDY, MD/PhD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No